CLINICAL TRIAL: NCT01091415
Title: Comparison of Volar Locking Plate Fixation Alone and Volar Locking Plate Fixation Plus Calcium Phosphate Bone Cement Augmentation for Distal Radius Fractures Patients Aged More Than 65
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Jae Kwang Kim, Ewha Womans Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECT
Record Dates: First submitted 2010-03-19; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-12

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- calcium phosphate bone cement (Experimental): one arm; volar locking plate alone the other arm; calcium phosphate bone cement as well as volar locking plate
  Interventions: Procedure: calcium phosphate bone cement injection

INTERVENTIONS:
Procedure: calcium phosphate bone cement injection — volar locking plate alone versus calcium phosphate bone cement as well as volar locking plate

SUMMARY:
The incidence of distal radius fracture (DRF) increases with age, and thus, because of improving life expectancies, these fractures are set to become more common. Fractures of the distal radial metaphysis are known to be strongly related to osteoporosis, and as a result, the management of distal radius fractures in elderly patients is beset with difficulties.

Recently, more aggressive fracture fixation in the elderly has become a topic of interest, in the hope of increasing the rate of recovery to preserve the ability to live independently. Many elderly patients remain active well into their eighth and ninth decades, for example, some pursue activities, such as, golf and tennis, on a daily basis. The introduction of volar locking plating system has increased this interest. This system, which uses a fixed angle principle, has been proposed to be effective at maintaining good anatomic reduction, even in the elderly. However, there is a still concern about remaining metaphyseal defect after reduction of the osteoporotic DRF.

Injectable calcium phosphate bone cement (CPC) has been used to augment the remaining metaphyseal defect after fracture reduction including DRF, specially in osteoporotic old patients. The purpose of this randomized, prospective study was to investigate that additional CPC augmentation has any benefit over volar locking plate fixation in unstable DRF patient who is older than 65. The null hypothesis is that there is no difference of wrist functional outcomes, radiographic outcomes, and complications between treatment of volar locking plate alone and calcium phosphate bone cement as well as volar locking plate in unstable DRF patient who is older than 65.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 65 years old with an acute DRF were considered for inclusion for this study. Inclusion criterion of this study was an unacceptable closed reduction after one attempt of closed reduction. The criteria of unacceptable closed reduction included dorsal angulation of > 100, volar angulation of > 200, an articular gap or step off of >2 mm, radial inclination of <100, or radial shortening of > 5mm.

Exclusion Criteria:

* A preexisting severe illness
* An ipsilateral upper extremity injury
* A previous wrist injury
* Surgical delay of more than 2 weeks
* A concomitant ulnar neck fracture.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | 12 months postoepratively
  grip strength, wrist range of motion, subjective wrist pain, modified Mayo wrist score, and Disabilities of Arm, Shoulder and Hand score

SECONDARY OUTCOMES:
Radiographic outcomes | postoperatively 12 months
  radial inclination and volar angulation and ulnar variance

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Orbay JL, Fernandez DL. Volar fixed-angle plate fixation for unstable distal radius fractures in the elderly patient. J Hand Surg Am. 2004 Jan;29(1):96-102. doi: 10.1016/j.jhsa.2003.09.015. PMID 14751111
- [Background] Larsson S, Bauer TW. Use of injectable calcium phosphate cement for fracture fixation: a review. Clin Orthop Relat Res. 2002 Feb;(395):23-32. doi: 10.1097/00003086-200202000-00004. PMID 11937863
- [Background] Ring D, Jupiter JB. Treatment of osteoporotic distal radius fractures. Osteoporos Int. 2005 Mar;16 Suppl 2:S80-4. doi: 10.1007/s00198-004-1808-x. Epub 2004 Dec 22. PMID 15614440